CLINICAL TRIAL: NCT04076826
Title: Adjunctive Sedation With Dexmedetomidine for the Prevention of Severe Inflammation and Septic Encephalopathy: a Pilot Randomized Controlled Study.
Brief Title: Adjunctive Sedation With Dexmedetomidine for the Prevention of Severe Inflammation and Septic Encephalopathy
Acronym: ADVISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Luca Cioccari, Dr. med., Insel Gruppe AG, University Hospital Bern
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4051
Record Dates: First submitted 2019-08-22; First posted 2019-09-03 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Sepsis-Associated Encephalopathy
Keywords: Sepsis; Dexmedetomidine; Sedation; S-100beta; Encephalopathy
MeSH Terms: conditions — Sepsis-Associated Encephalopathy; Sepsis; Brain Diseases | interventions — Dexmedetomidine; Propofol; Midazolam; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Protocol A (Dexmedetomidine) (Experimental): Dexmedetomidine will be administered in accordance with hospital standard operating procedures (SOP).
  Interventions: Drug: Dexmedetomidine; Diagnostic Test: Blood sampling
- Protocol B (Propofol / Midazolam) (Active Comparator): Propofol and/or Midazolam will be administered in accordance with hospital standard operating procedures (SOP).
  Interventions: Drug: Propofol or Midazolam; Diagnostic Test: Blood sampling

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine infusion will be commenced in accordance with the hospital's local sedation protocol, without a loading dose, at a rate of 0.1 - 1.4 mcg/kg/hour to maintain sedation as per Richmond Agitation-Sedation Scale (RASS) sedation range specified by the treating clinician. Infusion will be continued until sedation is no longer clinically indicated up to a maximum of 7 days after enrolment.
  Other Names: Protocol A
  Arms: Protocol A (Dexmedetomidine)
Drug: Propofol or Midazolam — Propofol and/or Midazolam will be used according to Hospital guidelines to maintain sedation as per Richmond Agitation-Sedation Scale (RASS) sedation range specified by the treating clinician.
  Other Names: Protocol B
  Arms: Protocol B (Propofol / Midazolam)
Diagnostic Test: Blood sampling — In all participants, we will collect blood samples for measurement of neuronal and systemic biomarkers of inflammation at randomization (baseline), at day 1, day 2 and day 3 after randomization.

SUMMARY:
Septic encephalopathy (SE) is defined as acute cerebral dysfunction in patients with sepsis or septic shock. SE occurs in up to 50% of critically ill patients with sepsis and is associated with a high mortality and morbidity. The pathophysiology of SE is complex and involves increased levels of inflammatory mediators such as tumor necrosis factor (TNF)-α, Interleukin (IL)-1 and IL-6, leading to blood brain barrier dysfunction and neuronal inflammation. Several biomarkers of neuronal injury have been proposed to identify patients with SE. Of these biomarkers, S100-β has the highest sensitivity and specificity.

Sedation with Dexmedetomidine (DEX) is a promising strategy for the management of these patients, as DEX has been shown to decrease the production of inflammatory mediators in experimental models of sepsis. In clinical studies, DEX lowers the incidence of delirium and critical illness polyneuropathy. However, its effectiveness in treatment and prevention of SE remains unclear.

The aim of the present study is to investigate the effect of two standard sedation protocols (Dexmedetomidine sedation vs. Propofol / Midazolam) on serum markers of SE in critically ill patients with sepsis who require sedation and mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* The participant is aged 18 years or older
* The participant has been intubated and is receiving mechanical ventilation
* The participant requires sedative medication for comfort, safety or to facilitate the delivery of life support measures
* The participant has either a central venous or an arterial catheter inserted within 24 hours of admission
* The participant has a diagnosis of sepsis based on the recent SEPSIS-3 consensus clinical criteria.

Exclusion Criteria:

* Age < 18 years
* The treating physician believes that the participant will remain intubated for <24 hours or the participant has been intubated for diagnostic or therapeutic procedures as the sole reason for mechanical ventilation.
* Participants with any of the following admission diagnosis: acute cerebral vascular event, traumatic brain injury, epilepsy, hypoxic brain injury, meningitis, encephalitis
* Participants with history of melanoma (S 100-β is elevated in melanoma participants)
* Participants with schizophrenia or other chronic psychiatric conditions
* Admission for drug overdose
* Planned administration of ongoing neuromuscular blockade
* Heart rate < 55 / min or an atrioventricular block > grade 2a in the absence of a functioning pacemaker
* Known hypersensitivity or allergy to any of the sedative medications used in this study.
* DNR (do not resuscitate) or DNI (do not intubate) orders
* Death is deemed to be imminent or inevitable during this admission and either the attending physician, participant or substitute decision maker is not committed to active treatment
* Women who are pregnant or breast feeding
* Known or suspected non-compliance, drug or severe alcohol abuse
* Inability of the participant to understand the procedures of the study, e.g. due to language problems, psychological disorders, or dementia
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
S100-ß | at 48 hours after randomization
  Serum concentration of S100-ß

SECONDARY OUTCOMES:
Neuron-specific enolase | first 3 days after randomization
  Serum concentration of Neuron-specific enolase
Interleukin 1-beta | first 3 days after randomization
  Serum concentration of Interleukin 1-beta
Interleukin 6 | first 3 days after randomization
  Serum concentration of Interleukin 6
TNF alpha | first 3 days after randomization
  Serum concentration of TNF alpha
Acetylcholinesterase activity | first 3 days after randomization
  Acetylcholinesterase activity will be measured using a point-of-care device and reported as Units/grams Haemoglobin
Butyrylcholinesterase activity | first 3 days after randomization
  Butyrylcholinesterase activity will be measured using a point-of-care device and reported as Units/L

CONTACTS AND LOCATIONS:
Overall Officials: Luca Cioccari, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iten M, Bachmann K, Jakob SM, Grandgirard D, Leib SL, Cioccari L. Adjunctive Sedation with Dexmedetomidine for the Prevention of Severe Inflammation and Septic Encephalopathy: A Pilot Randomized Controlled Study. Crit Care Med. 2025 Jul 1;53(7):e1377-e1388. doi: 10.1097/CCM.0000000000006655. Epub 2025 Mar 31. PMID 40162868